CLINICAL TRIAL: NCT03872492
Title: Major Depressive Disorder: Early Prediction of Non-response to Antidepressant Therapy Via a Mobile Digital Scale
Acronym: REDRESS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped prematurely because the total number of analyzable patients for the primary objective to be included was reached.
Sponsor: Ad scientiam (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: REDRESS
Record Dates: First submitted 2019-02-27; First posted 2019-03-13 (Actual); Last update posted 2023-03-03 (Actual); Status verified 2023-03

CONDITIONS: Depressive Disorder, Major
Keywords: REDRESS; Depression; Application; Mobile
MeSH Terms: conditions — Depressive Disorder, Major; Depression

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with Major Depressive Disorder (Experimental): Patients will be followed for 12 weeks. Hospital visits will be made at week 2 and week 6 (Phase1) as well as week 8 and week 12 (Phase 2).
  At the end of phase 1 if the patient is considered as an responder he will make one more visit at week 12.
  If the patient is considered as non-responder, he will make 2 other visits: at week 8 and week 12.
  Between each visit, the patient will perform REDRESS application assessments every day for "My daily survey" and every 3 days for the other assessments.
  Interventions: Other: Digital Assessment on mobile

INTERVENTIONS:
Other: Digital Assessment on mobile — The digital assessment is composed on 5 tests:
  * "My daily survey"
  * "My evaluation"
  * "My cognition"
  * "My emotions"
  * "My voice"
  Data will also be collected passively.

SUMMARY:
Major Depressive Disorder (MDD) is a debilitating disease characterized by a depressed mood, diminished interests, impaired cognitive function and vegetative symptoms, such as disturbed sleep or appetite. MDD occurs about twice as often in women than it does in men and affects about 6% of the adult population worldwide each year.

Standard symptoms scales like the Hamilton Depression Rating Scale or the Montgomery-asberg Depression Rating Scale, the Self-Report 16-item Quick Inventory of Depressive Symptomatology were initially developed for the evaluation of a therapeutic intervention or a pharmacological treatment and are routinely used by clinicians in the assessment of Treatment Resistant Depression (TRD) occurrence. In parallel, patient-reported outcomes have gained increasing importance and are widely recommended by health authorities in the assessment of depression. The same institutions insist on the collection of real-world data to provide clinicians with ecological measurements. It has been demonstrated that an early response to an AntiDepressant (AD) treatment can be seen as early as week 2 and is not related to a placebo-effect. While there is no consensus on the exact cut-off values, several factors emerge as early predictors of a later treatment response, such as:

* Improvement in emotional processing of happy facial expressions after 1 week of treatment,
* Circa 20% improvement in Hamilton Depression Rating Scale-17 item (HDRS-17) at week 2. The hypothesis is therefore that repeated, systematic and real-time, contextualized and multimodal collection of depressive symptoms from patients at home will establish a threshold score that can predict a subsequent response to their treatment.

REDRESS was inspired by several standard depression scales used and recommended by the French Health Authority, augmented with digital active and passive activity monitoring, speech analysis and emotional processing assessment. Another important assumption is that honesty and willingness to disclose personal or embarrassing things will be best achievable via a digital solution.

To test this assumption, the overall scores and each subscores on the REDRESS numerical scale will be compared in people with MDD showing adequate response to those showing insufficient response.

The response to treatment at week 6 will be studied (end of Phase 1). Non-responders and responders to the first treatment round will be enrolled in a 6-week extension phase (Phase 2). Non-responders will receive another treatment course (Other AD, combination, etc.). Responders will just be followed up and will keep the same treatment. The REDRESS scores will be analysed in this population and will allow us to test the investigator's assumption in people with treatment resistant depression. This study will also allow to assess patients' quality of life at the end of each phase of treatment and to compare results with REDRESS scores.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 70 Years
* Diagnostic and Statistical Manual of Mental Disorders-5 criteria for MDD
* Score > 21 on HDRS-17
* Initiation of an antidepressant treatment for the current episode (first line or second line treatment, ...)
* Ability to use a mobile application
* Agreement to use the study mobile if he/she does not own an iPhone 5 or newer
* Enrolled in or benefiting of a Social Security program
* Having read the information sheet and signed the informed consent form

Non inclusion Criteria:

* Serious suicidal risk, identified by the Mini International Neuropsychiatric Interview (MINI)
* Perinatal depression
* Seasonal affective disorder
* Psychiatric comorbidities: bipolar disorder, obsessive-compulsive disorder, post-traumatic stress, psychotic disorder, anorexia nervosa, bulimia nervosa, personality disorder identified by the MINI questionnaire
* Alcohol addiction or abuse, identified by the MINI questionnaire
* Substance related disorders non-alcoholic addiction or abuse (opioids, cocaine, cannabis, sedatives, stimulants, hallucinogens, inhalants, solvents), identified by the MINI questionnaire
* Under neurostimulation (< 6 months before inclusion day)
* Patient under Temporary Use Authorisation (TUA)
* Patients with Monoamine Oxidase Inhibitor (MAOIs), tricyclic antidepressant
* Patient with electroconvulsive therapy (ECT) history for current episode
* Patient with a somatic pathology
* Scheduled hospitalization for more than 7 days
* Antecedent of major head trauma
* Seizures
* Systemic medical diseases that are likely to affect cognitive functioning
* Pregnant and nursing women
* Wearers of pacemakers, implantable defibrillators
* Subjects not proficient in French
* Person under guardianship or curators
* Illiterate subjects
* Participation to another interventional clinical trial (category 1)

Exclusion criteria:

* Serious suicidal risk, according to clinician's judgement
* Discontinuation or change of AD treatment before 4 weeks after the dose initiation in the phase 1 and 2
* Initiation of a structured psychotherapy or neurostimulation
* Initiation of treatment with MAOIS
* Introduction of benzodiazepines at regular doses. Limited use (≤7 consecutive days or several periods of ≤3 consecutive days) is authorized
* Alcohol and substances abuse related disorders (opioids, cocaine, cannabis, sedatives, stimulants, hallucinogens, inhalants, solvents), according to clinician's judgement.
* Patient under Temporary Use Authorisation (TUA)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2019-10-17 (Actual); Primary Completion 2022-12-29 (Actual); Study Completion 2022-12-29 (Actual)

PRIMARY OUTCOMES:
Show that responders and non-responders in phase 1, have a different early profile on some of the items assessed by REDRESS at week 2 (or before) and identify the predictor item(s). | From Day 0 to Week 2
  Identification of items will be based on the diagnostic performance (AUC).

SECONDARY OUTCOMES:
Show that responders and non-responders in phase 1 have a different profile on some of the items assessed by REDRESS at week 6 and identify the discriminating item(s). | From Day 0 to Week 6
  Identification of items will be based on the diagnostic performance (AUC).
Reproducibility: show that responders and non-responders in phase 2 have a different profile on some of the items assessed by REDRESS at week 8 and identify the same predictor item(s) found in phase 1. | From Week 6 to Week 8
  Identification of items will be based on the diagnostic performance (AUC).
Reproducibility: show that responders and non-responders in phase 2 have a different profile on some of the items assessed by REDRESS at week 12 and identify the same discriminating item(s) found in phase 1. | From Week 6 to Week 12
  Identification of items will be based on the diagnostic performance (AUC).
Intra-patient comparison phase 1 / phase 2: show that patients non-responding in phase 1 and responding in phase 2 have a different profile on some of the items assessed by REDRESS | Between Week 6 and Week 12
  Intra patient comparison will be based on a paired comparison test.
Intra-patient comparison phase 1 / phase 2: show that patients non-responding in phase 1 and responding in phase 2 have a different profile on some of the items assessed by REDRESS | Between Week 2 and Week 8
  Intra patient comparison will be based on a paired comparison test.
Build up a composite score (the REDRESS digital score), from the item(s) identified in the previous objectives. | Week 2, Week 6, Week 8 and Week 12
  Ability of the REDRESS digital score to identify responders and non-responders will be based on the diagnostic performance.
  The REDRESS digital score will be built using the 5 assessments: "My Daily Survey", My Evaluation", "My Cognition", "My Emotion", My Voice" and passive data collection. This score will be constructed during the study.
Evaluate patients' adherence to the mobile application | From Day 0 to Week 12
  Patients' adherence to the REDRESS mobile application will be based on the number of questionnaires administered and completed and the number of variables collected via the mobile application as a function of time of follow-up.
Evaluate the adverse events of the mobile application use. | From Day 0 to Week 12
  Mobile application safety will be assessed by a descriptive analysis.
Collect patients and investigators feedback (usability, satisfaction) on the REDRESS mobile application | Week 12
  Descriptive analysis of patients and investigators satisfaction relating to the mobile application collected with satisfaction questionnaires
Evaluate patient's social relationship | Day 0, Week 6 and Week 12
  The quality of life will be measure with the form "Work and Social Adjustment Scale" (WSAS). This scale measures : ability to work, home management, social leisure activities, private leisure activities and close relationships. A WSAS score above 20 appears to suggest moderately severe or worse psychopathology. Scores between 10 and 20 are associated with significant functional impairment but less severe clinical symptomatology. Scores below 10 appears to be associated with subclinical populations. The maximum score of the WSAS is 40.
Evaluate patient's quality of life | Day 0, Week 6 and Week 12
  The quality of life will be measure with the form "Quality of Life Enjoyment". This questionnaire is designed to help assess the degree of enjoyment and satisfaction experienced during the past week. This scale mesures : physical health, mood, work, household activities, social relationship, family relationship, leisure time activities, ability to function in daily life, sexual drive, living situation, ability to do work or hobbies, medication.
Evaluate the patient's quality of life evolution | From Day 0 to Week 12
  The quality of life will be measure with the form "Work and Social Adjustment Scale" (WSAS). This scale measures : ability to work, home management, social leisure activities, private leisure activities and close relationships. A WSAS score above 20 appears to suggest moderately severe or worse psychopathology. Scores between 10 and 20 are associated with significant functional impairment but less severe clinical symptomatology. Scores below 10 appear to be associated with subclinical populations. The maximum score of the WSAS is 40.
Evaluate patient's social relationship evolution | From Day 0 to Week 12
  The quality of life will be measure with the form "Quality of Life Enjoyment". This questionnaire is designed to help assess the degree of enjoyment and satisfaction experienced during the past week. This scale mesures : physical health, mood, work, household activities, social relationship, family relationship, leisure time activities, ability to function in daily life, sexual drive, living situation, ability to do work or hobbies, medication.
Explore correlation between patient's quality of life and REDRESS score | Day 0, Week 6 and Week 12
  The correlation will be evaluated with the pearson correlation
Evaluate patient's quality of life | Day 0, Week 6 and Week 12
  The quality of life will be measure with the form "Dimensional Anhedonia Rating Scale". This scale measure anhedonia in the context of Major Depressive Disorder. The DARS assesses anhedonia across 4 domains: Hobbies, Food/Drink, Social Activities and Sensory Experiences.
  The total score of the DARS ranges from 0-68.

CONTACTS AND LOCATIONS:
Overall Officials: Bruno MILLET, Prof, Principal Investigator — Pitié-Salpêtrière Hospital
Locations (10):
- France (10):
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Grenoble, Grenoble
  - CHU Nantes - CAPPA Jacques Prévet, Nantes
  - CHU de Nice, Nice
  - Centre hospitalier Saint-Antoine, Paris
  - Hôpital de la Pitié Salpêtrière, Paris
  - Centre hospitalier Henri Laborit, Poitiers
  - Centre Hospitalier Guillaume Régnier, Rennes
  - CHU Toulouse, Toulouse
  - CHRU Tours, Tours